CLINICAL TRIAL: NCT04407637
Title: Kinematic Axial Cervical Rotation Performance in Patients With Acute Non-specific Neck Pain During the DidRen Laser Test is Improved After Passive Manual Cervical Mobilizations Regardless of the Painful Spinal Level
Brief Title: Kinematic Cervical Rotation Performance in Neck Pain Patients is Improved After Cervical Treatment
Acronym: DidRen
Status: Completed | Type: Observational
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Detrembleur, Professor, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Other Study IDs: RH_05_13_20
Record Dates: First submitted 2020-05-14; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Neck Pain
Keywords: fast neck rotation; sensorimotor control assessment
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- neck pain patients: Patients with acute non-specific neck pain were consecutively recruited from a private manual physiotherapy center as sample of convenience. Inclusion criteria were acute (<3months) non-specific neck pain with a neck disability index (NDI) > 8% and a Numerical Pain Rating Scale (NPRS) >3 . Patients were excluded if they reported any of the following: a history of neck surgery, dizziness caused by neck or head movements and cervical radiculopathy diagnosed by a physician.
- healthy: Healthy control participants were included if they reported a NDI < 8% and a NPRS =0. They were excluded if they reported neck pain during the last year, radiating symptoms in the shoulder or arm regions, or headache. Participants with a history of neck trauma or in treatment for spinal disorders or reporting pain during the manual assessment were excluded as well.

SUMMARY:
A longitudinal study is designed to assess the influence of acute non-specific neck pain on kinematic parameters during a fast-head axial rotation task standardized with the DidRen laser test device. First, the investigators will compare kinematic parameters between patients and healthy control. Second, the investigators will assess whether neck upper or lower pain location influenced kinematic parameters. Finally, the investigators will examine the short-term effect of passive cervical mobilizations in patients on these kinematic variables.

DETAILED DESCRIPTION:
At baseline, all participants will be asked to fill in four questionnaires.

* The Neck Disability Index (NDI), which is a self-rated instrument assessing disability due to neck pain, which consist of a series of 10 questions on activities relating to daily living all assessed on a 6-point scale.
* The Numerical Pain Rating Scale (NPRS), to assess the current neck pain.
* The Tampa scale of kinesiophobia (TSK), which is a 17-item questionnaire used to assess fear of movement or re-injury, in which participants are asked to rate their level of agreement with each item on a 1 (strongly disagree) to 4 (strongly agree) scale. The TSK has been shown to have adequate internal consistency (coefficient alpha 0.77) and to be associated with measures of behavioral avoidance and self-reported disability.A cut-off score above 39 is associated with a risk for prolonged pain-related disability.
* The French version of the Bournemouth Questionnaire based on the biopsychosocial model to evaluate different dimensions in neck pain participant including the pain, disability, affective and cognitive aspects of neck pain.

The investigators will assess the Fast Neck Rotation with the DidRen Test:

Also, clinical examination will include Cervical Rotation Testing, Manual Spinal Examination.

* The Didren laser test will be performed by the participant. During the DidRen Laser test, the kinematic rotation will be recorded using a validated Inertial Motion Unit (IMU). After the DidRen test, participant will rate their pain using the NPRS in order to assess if the pain intensity could interfere with the test performance.
* Measurements of cervical Rotation active range of motion (ROM) will be measured by an IMU. During active cervical ROM measurement participants will be asked to report any familiar pain on a Numerical Pain Rating Scale (NPRS). If no pain during active movement is reported, then the physiotherapist will passively move the head toward end of the ROM and note any stiffness and/or reported familiar pain from the participants. A positive cervical Rotation ROM test will be defined as the reproduction of stiffness and/or familiar cervical spine pain during the active ROM without or with over pressure.
* The Manual spinal examination will include Passive Physiological Intervertebral Movements (PPIVM's) in lateral flexion and extension and Passive Accessory Intervertebral Movements (PAIVM's), will be performed to detect the presence or absence of cervical joint dysfunction and to detect the region of the dysfunction either on the upper or lower region.The participant will be positioned supine for the PPIVM's and prone for the PAIVM's. For the PAIVM's, the assessor will apply centrally directed posterior-anterior (central P/A) force toward the spinous process or posterior-anterior directed force to the articular pillars (unilateral P/A) from the upper cervical region C0-1, C1-2 and C2-3 to the lower region C6-7 on each side. Any perceived resistance to passive motion will be recorded. The participant will be asked to report any familiar pain provocation on an NPRS. A positive test at a cervical level will be defined as a report of familiar local or referred pain when the assessor rate resistance to passive motion (Manual Spinal examination test have demonstrated moderate to excellent intrarater and interrater reliability in patients with axial neck pain referred for diagnostic facet joint blocks).

On the basis of the findings of the region of pain, subjects will enter either in the upper or lower cervical region group.

Regular baseline on the fast-head rotation task strategies standardized with the "DidRen Laser" device will be done by analyzing data from a control group constituted by asymptomatic subjects. As Manual Spinal Examination (P/A) has showed more sensitivity than specificity, asymptomatic subjects will also be excluded by the second assessor if during cervical Rotation ROM testing procedure and/or cervical manual examination.

Evaluation of Rotation ROM, Spinal Examination and first DidRen Test, will have already been completed.

The participant's treatment will include P/A mobilization . After treatment, Cervical ROM testing and the assessment of the fast Neck Rotation with the DidRen Test will be undergone by the participant:

The Therapist will apply PPIVM's at the symptomatic levels or PAIVM's either central posterior-anterior (central P/A) directed force toward the spinous process ora posterior-anterior directed force directed to the articular pillars (unilateral P/A) on spinal level(s) which were primary recorded as painful sites during the first spinal examination and referred to as "primary painful sites". As a treatment, Maitland Grade 3 and 4 will be used for the joint(s) mobilization(s) and could be performed at others symptomatic levels (these levels will be referred to as "secondary painful sites") depending on the subject's condition (which also contributes to reproduce familiar pain and /or stiffness). During treatment, the Musculoskeletal Physiotherapist will note all cervical levels mobilized, time and grades of movement used. The decision of the end of the treatment will be decided with minimal clinically important improvement (MCI) in pain and in disability. The MCI in pain is defined as a decrease by at least 2 points in pain intensity score at follow-up compared to baseline. The MCI in disability was defined as a decrease by at least 1 point in pain related disability (ROM) score at follow-up compared to baseline.

Assessment of cervical ROM (active + over pressure) by the IMU.The treatment will be performed a second time if no change occurs (MCI disability) after the first manual spinal treatment.

Assessment by the Didren laser test will be performed by the participant. After the DidRen test, participants will complete NPRS, in order to assess if the pain intensity could interfere with the performance of the test.

Musculoskeletal experience. · For blinding purposes, a second assessor will complete the DidRen Laser test.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Inclusion criteria were acute (<3months) non-specific neck pain with a neck disability index (NDI) > 8% and a Numerical Pain Rating Scale (NPRS) >3.
* Healthy control participants were included if they reported a NDI < 8% and a NPRS =0. They were excluded if they reported neck pain during the last year, radiating symptoms in the shoulder or arm regions, or headache. Participants with a history of neck trauma or in treatment for spinal disorders or reporting pain during the manual assessment were excluded as well.

Exclusion Criteria:

* Patients were excluded if they reported any of the following: a history of neck surgery, dizziness caused by neck or head movements and cervical radiculopathy diagnosed by a physician.
* Healthy: They were excluded if they reported neck pain during the last year, radiating symptoms in the shoulder or arm regions, or headache. Participants with a history of neck trauma or in treatment for spinal disorders or reporting pain during the manual assessment were excluded as well.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with acute non-specific neck pain were consecutively recruited from a private manual physiotherapy center as sample of convenience. Healthy were recruited from student population.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-02-02 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Change of head rotational speed (in °s-1) | T0: Before treatment; T1: after 6 weeks
  The head rotational speed (°s-1) was recorded using an inertial motion unit sensor. DYSKIMOT is an Ultra-Low-Cost Inertial Sensor to Assess Head's Rotational Kinematics in Adults during the Didren-Laser Test.
Change of head rotational acceleration (in °s-2) | T0: Before treatment; T1: after 6 weeks
  The head rotational acceleration (°s-2) was recorded using an inertial motion unit sensor. DYSKIMOT is an Ultra-Low-Cost Inertial Sensor to Assess Head's Rotational Kinematics in Adults during the Didren-Laser Test.
Change of head angular displacement (in °) | T0: Before treatment; T1: after 6 weeks
  The head angular displacement (°) was recorded using an inertial motion unit sensor. The DYSKIMOT is an Ultra-Low-Cost Inertial Sensor to Assess Head's Rotational Kinematics in Adults during the Didren-Laser Test.

SECONDARY OUTCOMES:
Change of Numerical Pain Rating Scale (NPRS). | T0: Before treatment; T1: after 6 weeks
  The Numerical Pain Rating Scale (NPRS) is a commonly used outcome to assess patients with neck pain. It uses an 11-point scale, ranging from 0 (no pain) to 10 (worst pain imaginable)

CONTACTS AND LOCATIONS:
Overall Officials: Christine Detrembleur, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Detrembleur, Brussels, Belgium

REFERENCES:
- [Derived] Hage R, Detrembleur C, Dierick F, Brismee JM, Roussel N, Pitance L. Sensorimotor performance in acute-subacute non-specific neck pain: a non-randomized prospective clinical trial with intervention. BMC Musculoskelet Disord. 2021 Dec 4;22(1):1017. doi: 10.1186/s12891-021-04876-4. PMID 34863120